CLINICAL TRIAL: NCT02194647
Title: Anti-osteoporosis Medication Monitoring and Management Service
Status: Active, not recruiting | Type: Observational
Sponsor: National Taiwan University Hospital (Other)
Responsible Party: Sponsor
Other Study IDs: 201406077RINA
Record Dates: First submitted 2014-07-16; First posted 2014-07-18 (Estimated); Last update posted 2024-09-20 (Actual); Status verified 2024-09

CONDITIONS: Osteoporosis; Fracture
Keywords: Osteoporosis; Medication Monitoring; Education; Adherence; Management
MeSH Terms: conditions — Osteoporosis; Fractures, Bone

STUDY DESIGN:
Observational Model: Case-Only | Time Perspective: Other
Oversight: Data Monitoring Committee: No

SUMMARY:
BACKGROUND:

One-year adherence to oral anti-osteoporosis medication (AOMs) was only about 30%. In recent years, efforts have been made to change the delivery of these medications from oral form to injection form every, 3, 6 or 12 months to increase adherence. However, both patients and providers are sometimes confused about the multiple choices. Also, patients may receive extra medications if providers did not keep tract of their previous AOM uses or patients may changes providers. There were urgent needs to provide AOM monitoring and management services to improve cares.

OBJECTIVES:

To establish a anti-osteoporosis medication management service at National Taiwan University Hospital and its BeiHu Branch.

METHODS:

Participating physicians will select those eligible for services and refer to study coordinators. Study coordinators will conduct baseline assessments on osteoporosis/fracture risks, record medical conditions, AOMs, provide educations on osteoporosis, fracture, sarcopenia, fall, medications, nutrition, and exercise. They also arrange return clinic visit, telephone reminder and follow up for patients, and communicate with providers on regular bases. the investigators plan to enroll 500 patients with 18-month follow up for each.

ELIGIBILITY:
Inclusion Criteria:

* Age >=50 and one of the below
* Newly prescribed with AOMs
* Recent change of AOMs
* Poor adherence to AOMs
* Participating physicians feel that the service will benefit the patient in overall osteoporosis and medication managements.

Exclusion Criteria:

* Life expectancy less than 2 years or can't be assessed for communication problems
* patient in our fracture liaison service or other medication clinical trials

Min Age: 50 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Adults treated with anti-osteoporosis medicines (AOMs)
Sampling Method: Non-Probability Sample
Enrollment: 500 (Actual)
Dates: Start 2014-07 (Actual); Primary Completion 2015-08-22 (Actual); Study Completion 2026-07-01 (Estimated)

PRIMARY OUTCOMES:
medication adherence | 18 months
  Medication adherence will be assessed at 4, 8, 12, 18 months after enrollments. Final results will be reported at 18 month. If the patient changes medication, all AOMs adherence will be combined.
  Specific formula is as below:
  for oral medications, adherence is defined as # medication taken/ #medication prescribed within past 3 months for injection medications, adherence is defined as # of injection/ # of due injection since baseline or last follow up phone call.
  Statistics: Simple counts of adherence % among all participants.

CONTACTS AND LOCATIONS:
Overall Officials: Ding-Cheng Chan, MD, PhD, Principal Investigator — National Taiwan University Hospital
Locations (1):
- National Taiwan University Hospital, Taipei, Taiwan